CLINICAL TRIAL: NCT01347073
Title: A Switch-Over, Open-Label Study of the Safety, Pharmacokinetics, and Efficacy of HPN-100, Followed by Long-Term Treatment With HPN-100, in Pediatric Subjects Under 6 Years of Age With Urea Cycle Disorders (UCDs)
Brief Title: Study of the Safety, Pharmacokinetics and Efficacy of HPN-100, in Pediatric Subjects With Urea Cycle Disorders (UCDs)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPN-100-012
Record Dates: First submitted 2011-04-29; First posted 2011-05-04 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Urea Cycle Disorders
Keywords: Urea Cycle Disorder; UCD; GT4P; Buphenyl; hyperammonemia; sodium phenylbutyrate
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Hyperammonemia | interventions — glycerol phenylbutyrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HPN-100 (Experimental): Switch over from sodium phenylbutyrate to open label HPN-100 oral liquid over 10 days then open label, long term treatment for 12 months
  Interventions: Drug: HPN-100

INTERVENTIONS:
Drug: HPN-100 — HPN-100 is a pro-drug of PAA that combines with glutamine to provide an alternative vehicle for waste nitrogen elimination. It is a liquid with minimal taste and odor. Approximately three teaspoons of HPN-100 (~17.4 mL) delivers an equivalent amount as PBA that 40 tablets of NaPBA.
  Other Names: RAVICTI; Glycerol phenylbuterate

SUMMARY:
This non-randomized, open-label study was approximately one year in duration and consisted of a short term NaPBA to HPN-100 switchover part involving two overnight stays followed by a 12-month long term treatment period involving monthly visits.

DETAILED DESCRIPTION:
This was an open-label study consisting of a 10-day switch-over period during which subjects were switched from their prescribed dose of sodium phenylbutyrate (BUPHENYLTM or NaPBA) to a dose of HPN-100 that delivered the same amount of the active ingredient, PBA, followed by long-term treatment with HPN-100 for up to 12 months. The study was designed to capture information important for evaluating safety, Pharmacokinetics, and efficacy while recognizing sampling limitations in young children and current standard of care. Patients eligible for this study included pediatric patients from 29 days to < 6 years of age with either a diagnosed or clinically suspected Urea Cycle Disorders (UCD) who are receiving a stable dose of the powder formulation of NaPBA. Subjects were clinically stable and had been receiving a stable dose NaPBA powder for at least 5 days at the time of enrollment.

During the switch-over part of the study, subjects switched from NaPBA to HPN-100 in one step and had two overnight stays with 24 hour blood sampling, the first of which was on Day 1, while still taking NaPBA, and the second of which was on approximately Day 10 while taking HPN-100. Subjects then continued in the long-term treatment phase which was 12 months in duration.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 29 days to < 6 years old. If the subject is born prematurely, calculation of the lower age limit begins at the corrected gestational age of 40 weeks.
* Signed informed consent by the subject's legally acceptable representative
* Suspected or confirmed UCD diagnosis of any subtype, except NAGS deficiency
* On stable dose of NaPBA powder for at least 5 days before Day 1
* Not receiving sodium benzoate for at least 5 days before Day 1
* No concomitant illness which would preclude safe participation as judged by the investigator
* Able to receive medication orally
* Has not undergone liver transplantation, including hepatocellular transplantation
* Judged sufficiently stable and compliant with diet and treatment to be suitable for enrollment

Exclusion Criteria:

* Screening ammonia level > 100 μmol/L and signs and symptoms indicative of hyperammonemia; subjects may be rescreened after their ammonia is controlled and they are clinically stable, at the discretion of the investigator
* Use of any investigational drug within 30 days of Day 1
* Active infection (viral or bacterial) or any other condition that may increase ammonia levels
* Any clinical or laboratory abnormality of Grade 3 or greater severity according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.03, except Grade 3 elevations in ammonia and liver enzymes, defined as levels 5-20 times ULN (upper limit of normal)in alanine aminotransferase (ALT), aspartate aminotransferase (AST), or gamma glutamyl transpeptidase (GGT) in a clinically stable subject
* Any clinical or laboratory abnormality or medical condition that, at the discretion of the investigator, may put the subject at increased risk by participating in this study
* Known hypersensitivity to PAA or PBA
* Liver transplant, including hepatocellular transplant
* Currently treated with Carbaglu® (carglumic acid)

Ages: 29 Days to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2011-07; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: F MD, Study Director — Amgen
Locations (8):
- United States (8):
  - UCLA Pediatrics/Genetics, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Maine Medical Center, Portland, Maine
  - University of Minnesota, Minneapolis, Minnesota
  - Mount Sinai School of Medicine, New York, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Mokhtarani M, Diaz GA, Rhead W, Berry SA, Lichter-Konecki U, Feigenbaum A, Schulze A, Longo N, Bartley J, Berquist W, Gallagher R, Smith W, McCandless SE, Harding C, Rockey DC, Vierling JM, Mantry P, Ghabril M, Brown RS Jr, Dickinson K, Moors T, Norris C, Coakley D, Milikien DA, Nagamani SC, Lemons C, Lee B, Scharschmidt BF. Elevated phenylacetic acid levels do not correlate with adverse events in patients with urea cycle disorders or hepatic encephalopathy and can be predicted based on the plasma PAA to PAGN ratio. Mol Genet Metab. 2013 Dec;110(4):446-53. doi: 10.1016/j.ymgme.2013.09.017. Epub 2013 Oct 8. PMID 24144944
- [Derived] Smith W, Diaz GA, Lichter-Konecki U, Berry SA, Harding CO, McCandless SE, LeMons C, Mauney J, Dickinson K, Coakley DF, Moors T, Mokhtarani M, Scharschmidt BF, Lee B. Ammonia control in children ages 2 months through 5 years with urea cycle disorders: comparison of sodium phenylbutyrate and glycerol phenylbutyrate. J Pediatr. 2013 Jun;162(6):1228-34, 1234.e1. doi: 10.1016/j.jpeds.2012.11.084. Epub 2013 Jan 13. PMID 23324524

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Locations: Houston, TX; Minneapolis, MN; Washington, DC; New York, NY; Cleveland, OH; Portland, ME; Portland, OR
  Study Initiation Date: September 9, 2011 Study Completion Date: April 4, 2013
Pre-assignment Details: This is an open-label, fixed-sequence NaPBA to HPN-100 switchover study with no control group.
Groups:
- HPN-100: The first part of this open-label study consisted of a switch-over period during which patients were switched from the current medication (NaPBA) to HPN-100. The second part of this open-label study consisted of a 12-month long-term treatment phase with HPN-100. All participants in the switch-over were enrolled into the long-term treatment phase.
Period: Overall Study
Arm/Group | HPN-100
Started | 23
Completed | 21
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Liver Transplant | 1

BASELINE CHARACTERISTICS:
Population: Analyses were based on the safety population, defined as all patients who received any amount of study medication.
Arm/Group | HPN-100
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Rate of adverse events during the Switch-Over portion of the Protocol
Time Frame: 2 weeks
Population: All patients who received any amount of study medication were included in this population, which is the primary population for all baseline, accountability, demographic and safety analyses.
Measure: Number; unit: participants
Groups:
- NaPBA: Switch Over Arm
- HPN-100: Switch Over and Long Term Treatment Arm
Arm/Group | NaPBA | HPN-100
Number analyzed (Participants) | 15 | 15
participants | 0 | 6

2. Secondary Outcome: Blood Ammonia
Description: 24-hour ammonia AUC of blood ammonia levels on Days 1 (NaPBA) and 10 (HPN-100) were compared. Ammonia was assessed at Hour 0 (pre-first dose, fasted), Hour 8 (~2-4 hours after lunch or the second main meal and dose of NaPBA), Hour 12 (~4 hours after the last main meal) and 24 hours post-first dose (pre-first dose on following day, fasted).
Time Frame: 2 weeks
Population: All patients who received any amount of both study medications (NaPBA and HPN-100) were included in this population, which is the primary population for analysis of efficacy and pharmacokinetic parameters.
Measure: Mean (Standard Deviation); unit: umol/L*hours
Groups:
- NaPBA: Switch Over
- HPN-100: Switch Over and Long Term Treatment
Arm/Group | NaPBA | HPN-100
Number analyzed (Participants) | 15 | 15
umol/L*hours | 914.43 (630.21) | 647.63 (379.94)

3. Secondary Outcome: Frequency of Ammonia Levels Greater Than the Upper Limit of Normal (ULN) on HPN-100 Compared With NaPBA
Description: Ammonia values were converted to SI units (umol/L) and normalized to a standard ULN of 35 umol/L prior to analysis
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Number; unit: Ammonia Values > ULN
Units Other Than Participants: Ammonia Values
Arm/Group | NaPBA | HPN-100
Number analyzed (Participants) | 15 | 15
Number analyzed (Ammonia Values) | 58 | 53
Ammonia Values > ULN | 22 | 8

4. Secondary Outcome: Hyperammonemic Crisis
Description: Rate of HAC during pre-enrollment on NaPBA compared to HAC during HPN-100 treatment
Time Frame: 1 year
Measure: Number; unit: number of crises
Groups:
- Pre-enrollment: 12-months preceding the study
- Long-term Phase: The second part of this open-label study consisted of a 12-month long-term treatment phase with HPN-100. All participants in the switch-over were enrolled into the long-term treatment phase.
Arm/Group | Pre-enrollment | Long-term Phase
Number analyzed (Participants) | 23 | 23
number of crises | 29 | 12

5. Primary Outcome: Adverse Events
Description: Rate of adverse events during the Safety Extension portion of the protocol ( please note: HPN-100 treatment only during Safety Extension )
Time Frame: 12 months
Population: All patients that entered the Safety Extension were included in the analysis of adverse events
Measure: Number; unit: participants
Groups:
- HPN-100: Long Term Treatment
Arm/Group | HPN-100
Number analyzed (Participants) | 23
participants | 23

ADVERSE EVENTS:
Time Frame: Approximately 1 year, 7 months (from study initiation date to 30 days after study completion date)
Arm/Group | HPN-100
Serious Adverse Events (participants affected / at risk) | 11/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HPN-100 (N=23)
Hyperammonemia (Metabolism and nutrition disorders) | 7
Vomiting (Gastrointestinal disorders) | 2
Convulsion (Nervous system disorders) | 2
Gastroenteritis (Gastrointestinal disorders) | 1
Chemical Burn (Injury, poisoning and procedural complications) | 1
Hypophagia (Metabolism and nutrition disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HPN-100 (N=23)
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Diarrhea (Gastrointestinal disorders) | 6
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 12
Pyrexia (General disorders) | 9
Ear infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 4
Otitis media (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 14
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood bicarbonate decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 3
Hyperammonemia (Metabolism and nutrition disorders) | 7
Hypophagia (Metabolism and nutrition disorders) | 2
Convulsion (Nervous system disorders) | 2
Hyporeflexia (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4
Rash papular (Skin and subcutaneous tissue disorders) | 3
Skin odor abnormal (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
The protocol was designed to capture information important for evaluating safety, pharmacokinetics, and efficacy while recognizing sampling limitations in young children and current standard of care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No